CLINICAL TRIAL: NCT00833833
Title: A Phase I/II Multicenter, Randomized, Open Label, Dose-Escalation Study To Determine The Maximum Tolerated Dose, Safety, And Efficacy Of CC-4047 Alone Or In Combination With Low-Dose Dexamethasone In Patients Wth Relapsed And Refractory Multiple Myeloma Who Have Received Prior Treatment That Includes Lenalidomide And Bortezomib
Brief Title: MTD, Safety, and Efficacy of Pomalidomide (CC-4047) Alone or With Low-dose Dexamethasone in Patients With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-002
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone; dexamethasone 21-phosphate; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1: 2 mg pomalidomide (Experimental): Pomalidomide 2 mg daily on days 1-21 of each 28-day cycle. Participants with progressive disease (PD) had the option of adding dexamethasone 40 mg on Days 1, 8, 15, 22 of each 28-day cycle to the pomalidomide treatment, or discontinuing study treatment.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin
- Phase 1: 3 mg pomalidomide (Experimental): Pomalidomide 3 mg daily on days 1-21 of each 28-day cycle. Participants with progressive disease (PD) had the option of adding dexamethasone 40 mg on Days 1, 8, 15, 22 of each 28-day cycle to the pomalidomide treatment, or discontinuing study treatment.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin
- Phase 1: 4 mg pomalidomide (Experimental): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Participants with progressive disease (PD) had the option of adding dexamethasone 40 mg on Days 1, 8, 15, 22 of each 28-day cycle to the pomalidomide treatment, or discontinuing study treatment.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin
- Phase 1: 5 mg pomalidomide (Experimental): Pomalidomide 5 mg daily on days 1-21 of each 28-day cycle. Participants with progressive disease (PD) had the option of adding dexamethasone 40 mg on Days 1, 8, 15, 22 of each 28-day cycle to the pomalidomide treatment, or discontinuing study treatment.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin
- Phase 2: pomalidomide + dexamethasone (Experimental): Combination therapy of 4 mg pomalidomide given once per day on Days 1-21 of each 28-day cycle and the starting dose of dexamethasone (determined by age) on days 1, 8, 15, and 22 of each 28-day cycle. The starting dose of dexamethasone was 40 mg for participants who were ≤ 75 years of age and 20 mg for participants who were > 75 years of age. Dose reduction steps for dexamethasone were provided for drug-related toxicities.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin
- Phase 2: pomalidomide (Experimental): 4 mg pomalidomide was given once per day on Days 1-21 of each 28-day cycle until PD. Participants in the single agent pomalidomide treatment arm who developed confirmed PD at any time had the option to receive oral dexamethasone on days 1, 8, 15, and 22 of each 28-day cycle at the starting dose of 20 or 40 mg depending on age in addition to their current dose of pomalidomide, or to discontinue treatment.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Aspirin

INTERVENTIONS:
Drug: Pomalidomide — 1 mg, 2 mg, and 5 mg capsules for oral administration packaged in bottles containing a 21-day supply
  Other Names: CC-4047; Pomalyst
Drug: Dexamethasone — oral dexamethasone
  Other Names: dexamethasone sodium phosphate
Drug: Aspirin — As prophylactic anti-thrombotic treatment, all participants were given aspirin 81-100 mg daily (commercial supply) unless contraindicated. If aspirin was contraindicated, participants were given another form of anti-thrombotic therapy according to hospital guidelines or physician preference.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and effectiveness of the study drug (CC-4047) Alone Or in Combination With Low-dose Dexamethasone as treatment for patients with relapsed and refractory multiple myeloma

DETAILED DESCRIPTION:
The Phase 1 segment of the study was designed to determine the maximum tolerated dose (MTD) of single-agent pomalidomide, which was to be determined in the first cycle of treatment. Following completion of the first cycle, participants were allowed to continue the study at their assigned dose of pomalidomide.

Participants who developed progressive disease (PD) at any time, or who had not achieved at least a 25% reduction of serum myeloma (M)-protein levels (if measurable) and a 50% reduction of urine M-protein (if measurable) compared with baseline after completion of 4 cycles of pomalidomide, had the option to receive oral dexamethasone 40 mg on days 1, 8, 15, and 22 of each 28-day treatment cycle in addition to their current dose of pomalidomide. Participants with PD who chose not to add dexamethasone to pomalidomide therapy were to be discontinued from the study. Participants who chose to add dexamethasone were allowed to continue study treatment until PD developed again, unacceptable toxicity or participant withdrew consent, at which time they were to be discontinued.

Based on results from the phase 1 portion, the Data Monitoring Committee confirmed 4 mg/day as MTD of pomalidomide. Therefore, the recommended starting dose of pomalidomide for Phase 2 was 4 mg/day on Days 1-21 of each 28-day cycle. In the combination treatment arm, the starting dose of dexamethasone was 40 mg once per day. For subjects who were > 75 years of age, the starting dose of dexamethasone was 20 mg once per day. To prevent blood clots, all participants were to be given aspirin 81-100 mg daily (commercial supply) unless contraindicated. If contraindicated, another form of anti-thrombotic therapy was provided.

Participants in the Phase II combination treatment arm could continue study treatment until PD developed, at which time they were to be discontinued. Participants in the single agent pomalidomide treatment arm who developed PD, confirmed by the IRAC, at any time had the option to receive oral dexamethasone in addition to their current dose of pomalidomide at the starting dose described above. Participants with PD who chose not to add dexamethasone to pomalidomide therapy were discontinued from study treatment. Participants who chose to add dexamethasone to pomalidomide therapy could continue study treatment until PD developed again, unacceptable toxicity or participant withdrew consent, at which point they were discontinued.

Upon discontinuation from study treatment for PD or any other reason, participants were to be assessed two times per year, up to five years, for survival, second primary malignancy and subsequent anti-myeloma therapies.

Two analyses were planned during the course of the Phase 2 segment: one interim analysis (at 50% information of progression-free survival (PFS) events) and one final analysis. The Data Monitoring Commmittee recommended that Celgene personnel be unblinded based on the strength of the data. Subsequently, Celgene decided to file an application based on more current study data. The product was approved by the FDA in February 2013.

Since no further analyses are required per protocol nor to support the marketing application, the study was amended to remove undue burden from patients who remain on active treatment by ending the treatment segments of this study and transferring all active patients tothe Long-term Follow-up Phase. These patients who continue to be treated with pomalidomide will be provided Pomalyst through the Celgene Patient Support Program (Pomalyst REMSTM) until disease progression, unacceptable toxicity, the investigator decides to change therapy or patient decision. Investigators will treat their patients according to the local standard of care and follow the assessments required for patients in the Long-term Follow-up Phase. These assessments include subsequent myeloma therapies, second primary malignancies and survival.

The study continues. A final analysis will be performed when the study is completed and results reported as available.

ELIGIBILITY:
Inclusion Criteria:

* Must be greater than or equal to 18 years at the time of signing the informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Have a documented diagnosis of multiple myeloma and have relapsed and refractory disease. Patients must have received at least 2 prior therapies. Patients must have relapsed after having achieved at least stable disease for at least one cycle of treatment to at least one prior regimen and then developed PD. Patients must also have documented evidence of PD during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry (refractory disease)
* Patients must have also undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of bortezomib (either in separate regimens or within the same regimen)
* Measurable levels of myeloma paraprotein in serum (greater than or equal to 0.5 g/dL) or urine (greater than or equal 0.2 g/dL excreted in a 24 hour collection sample)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Females of childbearing potential (FCBP) [An FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months)] must agree to refrain from becoming pregnant for 28 days prior to initiation of study drug, while on study drug and for 28 days after discontinuation of study drug and must agree to regular pregnancy testing during this timeframe.
* All patients must also agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study
* Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 28 days following discontinuation from this study even if he has undergone a successful vasectomy. Males must also agree to refrain from donating blood, semen or sperm during the above referenced timeframe.
* All patients must agree not to share medication with another person.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form.
* Any serious concurrent medical conditions that may make the patient non-evaluable or put the patient's safety at risk.
* Pregnant or lactating females
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1,000 cells/mm3
  * Platelet count < 75,000/mm3 for patients in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/mm3 for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
  * Serum creatinine > 3.0 mg/dL
  * Serum glutamic oxaloacetic transaminase/Aspartate transaminase (SGOT/AST) or Serum Glutamic Pyruvate Transaminase/Alanine transaminase (SGPT/ALT) > 3.0 X upper limit of normal (ULN)
  * Serum total bilirubin > 2.0 mg/dL
* Prior history of malignancies, other than multiple myeloma, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix or breast
  * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection
* Hypersensitivity to thalidomide, lenalidomide, or dexamethasone
* Peripheral neuropathy ≥ Grade 2
* Use of any anti-myeloma drug therapy within 14 days of the initiation of study drug treatment or use of any experimental non-drug therapy within 28 days of the initiation of study drug treatment
* Radiation therapy within 14 days of initiation of study drug treatment Inability or unwillingness to comply with birth control requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars A Sternas, MD, Study Director — Celgene Corporation
Locations (19):
- United States (14):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Mass General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer CenterDivision of Hematology/Oncology, Ann Arbor, Michigan
  - Mayo Clinic - Arizona, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute Department of Medicine, Buffalo, New York
  - Mt. Sinai Hospital, New York, New York
  - Ohio State University Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (5):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital and University of Toronto, Toronto, Ontario
  - Royal Victoria Hosptial, Montreal, Quebec

REFERENCES:
- [Derived] Siegel DS, Weisel KC, Dimopoulos MA, Baz R, Richardson P, Delforge M, Song KW, San Miguel JF, Moreau P, Goldschmidt H, Cavo M, Jagannath S, Yu X, Hong K, Sternas L, Zaki M, Palumbo A. Pomalidomide plus low-dose dexamethasone in patients with relapsed/refractory multiple myeloma and moderate renal impairment: a pooled analysis of three clinical trials. Leuk Lymphoma. 2016 Dec;57(12):2833-2838. doi: 10.1080/10428194.2016.1177181. Epub 2016 Jun 7. PMID 27267105
- [Derived] Richardson PG, Siegel DS, Vij R, Hofmeister CC, Baz R, Jagannath S, Chen C, Lonial S, Jakubowiak A, Bahlis N, Song K, Belch A, Raje N, Shustik C, Lentzsch S, Lacy M, Mikhael J, Matous J, Vesole D, Chen M, Zaki MH, Jacques C, Yu Z, Anderson KC. Pomalidomide alone or in combination with low-dose dexamethasone in relapsed and refractory multiple myeloma: a randomized phase 2 study. Blood. 2014 Mar 20;123(12):1826-32. doi: 10.1182/blood-2013-11-538835. Epub 2014 Jan 13. PMID 24421329
- [Derived] Richardson PG, Siegel D, Baz R, Kelley SL, Munshi NC, Laubach J, Sullivan D, Alsina M, Schlossman R, Ghobrial IM, Doss D, Loughney N, McBride L, Bilotti E, Anand P, Nardelli L, Wear S, Larkins G, Chen M, Zaki MH, Jacques C, Anderson KC. Phase 1 study of pomalidomide MTD, safety, and efficacy in patients with refractory multiple myeloma who have received lenalidomide and bortezomib. Blood. 2013 Mar 14;121(11):1961-7. doi: 10.1182/blood-2012-08-450742. Epub 2012 Dec 14. PMID 23243282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2: Participants were stratified by age (≤ 75 vs. > 75), prior number of treatments (2 vs. > 2), and prior thalidomide exposure (yes vs. no).
Groups:
- Phase 1: 2 mg Pomalidomide: Pomalidomide 2 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
- Phase 1: 3 mg Pomalidomide: Pomalidomide 3 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
- Phase 1: 4 mg Pomalidomide: Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
- Phase 1: 5 mg Pomalidomide: Pomalidomide 5 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
- Phase 2: Pomalidomide + Dexamethasone: Combination therapy of 4 mg pomalidomide given once per day on Days 1-21 of each 28-day cycle and the starting dose of dexamethasone (either 40mg or 20 mg) on days 1, 8, 15, and 22 of each 28-day cycle.
- Phase 2: Pomalidomide: 4 mg pomalidomide was given once per day on Days 1-21 of each 28-day cycle until PD. Participants in the single agent pomalidomide treatment arm who developed confirmed PD at any time had the option to receive oral dexamethasone at the starting dose in addition to their current dose of pomalidomide, or to discontinue treatment.
Period: Phase 1 (as of 01 April 2011)
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Started | 6 | 8 | 14 | 10 | 0 | 0
Completed | 2 (Confirmed progressive disease) | 3 (Confirmed progressive disease) | 5 (Confirmed progressive disease) | 4 (Confirmed progressive disease) | 0 | 0
Not Completed | 4 | 5 | 9 | 6 | 0 | 0
Not completed — Still active in study | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Disease progression - unconfirmed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 3 | 0 | 1 | 0 | 0
Period: Phase 2 (as of 01 April 2011)
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Started | 0 | 0 | 0 | 0 | 113 | 108
Safety Population | 0 | 0 | 0 | 0 | 112 | 107
Completed | 0 | 0 | 0 | 0 | 58 (Confirmed progressive disease) | 47 (Confirmed progressive disease)
Not Completed | 0 | 0 | 0 | 0 | 55 | 61
Not completed — Still active in study | 0 | 0 | 0 | 0 | 23 | 22
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 8 | 13
Not completed — Death | 0 | 0 | 0 | 0 | 8 | 9
Not completed — Disease progression - unconfirmed | 0 | 0 | 0 | 0 | 7 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 7
Not completed — Other | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population from both phases
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide | Total
Number analyzed (Participants) | 6 | 8 | 14 | 10 | 113 | 108 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.83) | 70.4 (6.63) | 67.5 (8.98) | 61.3 (14.06) | 64.4 (9.24) | 62.9 (10.35) | 64.1 (9.86)
Age, Customized [Number; unit: participants]
  <=75 years | 6 | 6 | 11 | 9 | 99 | 95 | 226
  >75 years | 0 | 2 | 3 | 1 | 14 | 13 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 6 | 51 | 51 | 122
  Male | 1 | 3 | 10 | 4 | 62 | 57 | 137
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 2 | 2 | 3 | 7
  Black or African American | 1 | 0 | 0 | 0 | 17 | 16 | 34
  White | 5 | 8 | 14 | 8 | 92 | 86 | 213
  Other | 0 | 0 | 0 | 0 | 2 | 3 | 5
Baseline Electrocardiogram Findings [Number; unit: participants]
  Normal | 3 | 3 | 3 | 4 | 53 | 44 | 110
  Abnormal, not clinically significant | 3 | 5 | 11 | 6 | 56 | 59 | 140
  Abnormal, clinically significant | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Missing | 0 | 0 | 0 | 0 | 4 | 4 | 8
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — The ECOG scale is as follows:
  Grade 0: Fully active, able to carry on all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair.
  participants
    0 | 1 | 0 | 3 | 2 | 32 | 24 | 62
    1 | 1 | 8 | 10 | 5 | 68 | 71 | 163
    2 | 4 | 0 | 1 | 3 | 13 | 11 | 32
    3 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Baseline Multiple Myeloma Stage [Number; unit: participants] — Multiple myeloma has three stages, which are known as stage I, stage II and stage III. Staging in myeloma is done on the basis of the value of serum albumin and beta-2 microglobulin level. Stage I has the best prognosis and stage III the worst prognosis.
  participants
    Stage I | 1 | 1 | 3 | 2 | 8 | 8 | 23
    Stage II | 0 | 1 | 4 | 1 | 29 | 29 | 64
    Stage III | 5 | 6 | 7 | 7 | 76 | 71 | 172
Prior Anti-Myeloma Therapies [Number; unit: participants]
  Yes | 6 | 8 | 14 | 10 | 113 | 108 | 259
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prior Thalidomide Exposure [Number; unit: participants]
  Yes | 4 | 6 | 11 | 9 | 76 | 72 | 178
  No | 2 | 2 | 3 | 1 | 37 | 36 | 81
Prior Stem Cell Transplant [Number; unit: participants]
  Yes | 4 | 4 | 11 | 6 | 84 | 82 | 191
  No | 2 | 4 | 3 | 4 | 29 | 26 | 68

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Participants With Dose-Limiting Toxicities (DLT) in Cycle 1
Description: The maximum tolerated dose was defined as the highest dose level at which no more than 1 of 6 participants experiences a DLT within the first 28-day cycle.
  DLTs were defined as:
  * Grade 4 neutropenia or thrombocytopenia
  * Febrile neutropenia
  * Grade 3 or 4 nausea, vomiting or diarrhea despite optimal symptomatic treatment
  * Serum transaminase > 20 * upper limit of normal (ULN)
  * Serum transaminase > 5 * ULN for >= 7 days
  * Delay of the start of cycle 2 by >7 days due to pomalidomide-related adverse event
Time Frame: Up to Day 28 (Cycle 1)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide
Number analyzed (Participants) | 6 | 8 | 14 | 10
participants | 1 | 1 | 2 | 4

2. Primary Outcome: Phase 2: Kaplan-Meier Estimates of Progression-free Survival (PFS) as of the 01 April 2011 Cut-off
Description: Progression free survival (PFS) is the time from randomization to the first documentation of disease progression or death from any cause during study, whichever occurs earlier. Disease progression was assessed by the Independent Response Adjudication Committee (IRAC).
  For the primary PFS analysis, participants who withdrew for any reason or received another antimyeloma therapy (except adding dexamethasone to the Phase 2: Pomalidomide arm) without documented PD (as determined by the IRAC review) were censored on the date of their last adequate response assessment, prior to receiving any other anti-myeloma therapy. Subjects who were still active at the time of the data cut-off date without PD (as determined by the IRAC) were censored on the date of their last adequate response assessment.
  Data collection is ongoing and future data results will be included as available.
Time Frame: up to 67 weeks
Population: Intent to treat population.
  Data collection is ongoing and future data results will be included as available.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 113 | 108
weeks | 16.6 [14.1 to 21.1] | 10.7 [8.3 to 16.1]
Statistical Analysis 1: Comparison: Phase 2: Pomalidomide + Dexamethasone vs Phase 2: Pomalidomide; With a 12-month accrual period and 12-month follow-up after the study closed to accrual, assuming a 10% drop out rate, 96 participants in each treatment arm would have had 85% power to detect a hazard rate ratio of 1.67 using a one-sided log rank test with an overall significance level of 0.025 adjusted for one interim analysis) and a significance level of 0.0245 for the final analysis; Test type: Superiority or Other; Cox Proportional Hazard = 0.73, 95% CI 2-sided [0.54 to 0.99]

3. Secondary Outcome: Phase 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) While on Single-Agent Pomalidomide as of the 01 April 2011 Cut-off
Description: Relation to study drug was assessed by the Investigator as either suspected or not suspected. Counts represent the suspected relationship. Severity was assessed using National Cancer Institute Common Toxicity Terminology Criteria for Adverse Events version 3.0 (NCI CTCAE v3.0): 1= Mild 2= Moderate 3= Severe 4= Life-threatening and 5= Death related to AE. Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
  Data collection is ongoing and future data results will be included as available.
Time Frame: Up to week 104
Population: Safety population.
  Data collection is ongoing and future data results will be included as available.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide
Number analyzed (Participants) | 6 | 8 | 14 | 10
percentage of participants
  1 or more (1+) AE | 100.0 | 100.0 | 100.0 | 100.0
  1+ AE related to pomalidomide | 66.7 | 75.0 | 85.7 | 100.0
  1+ severity grade 3-4 AE | 83.3 | 37.5 | 78.6 | 80.0
  1+ severity grade 3-4 AE related to pomalidomide | 33.3 | 25.0 | 42.9 | 70.0
  1+ serious AE (SAE) | 50.0 | 12.5 | 42.9 | 30.0
  1+ SAE related to pomalidomide | 0.0 | 12.5 | 7.1 | 10.0
  1+ AE leading to discontinuation of pomalidomide | 16.7 | 0.0 | 21.4 | 0.0
  1+AE-dose reduction/interruption of pomalidomide | 16.7 | 75.0 | 42.9 | 80.0
  1+related AE-reduction/interruption of pomalidomid | 0.0 | 37.5 | 28.6 | 70.0

4. Secondary Outcome: Phase 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) While on Both Pomalidomide and Dexamethasone as of the 01 April 2011 Cut-off
Description: TEAEs that occurred during Phase 1 after dexamethasone was added to pomalidomide treatment.
  Relation to study drug was assessed by the Investigator as either suspected or not suspected. Counts represent the suspected relationship. Severity was assessed using National Cancer Institute Common Toxicity Terminology Criteria for Adverse Events version 3.0 (NCI CTCAE v3.0): 1= Mild 2= Moderate 3= Severe 4= Life-threatening and 5= Death related to AE. Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
  Data collection is ongoing and future data results will be included as available.
Time Frame: Up to week 126
Population: Safety population.
  Data collection is ongoing and future data results will be included as available.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide
Number analyzed (Participants) | 1 | 4 | 10 | 7
percentage of participants
  1 or more (1+) AE | 100.0 | 100.0 | 90.0 | 100.0
  1+ AE related to pomalidomide | 100.0 | 75.0 | 80.0 | 100.0
  1+ AE related to dexamethasone | 100.0 | 75.0 | 70.0 | 85.7
  1+ severity grade 3-4 AE | 0.0 | 75.0 | 70.0 | 57.1
  1+ severity grade 3-4 AE related to pomalidomide | 0.0 | 75.0 | 20.0 | 42.9
  1+ severity grade 3-4 AE related to dexamethasone | 0.0 | 75.0 | 20.0 | 0.0
  1+ serious AE (SAE) | 0.0 | 75.0 | 40.0 | 28.6
  1+ SAE related to pomalidomide | 0.0 | 25.0 | 20.0 | 0.0
  1+ SAE related to dexamethasone | 0.0 | 50.0 | 10.0 | 0.0
  1+ AE leading to discontinuation of pomalidomide | 0.0 | 25.0 | 20.0 | 0.0
  1+ AE -- discontinuation of dexamethasone | 0.0 | 25.0 | 20.0 | 0.0
  1+AE -dose reduction/interruption of pomalidomide | 0.0 | 50.0 | 40.0 | 71.4
  1+ AE-dose reduction/interruption of dexamethasone | 0.0 | 75.0 | 60.0 | 71.4
  1+related AE-reduction/interruption of pomalidomid | 0.0 | 25.0 | 20.0 | 57.1
  1+related AE-reduction/interruption of dexamethaso | 0.0 | 75.0 | 20.0 | 42.9

5. Secondary Outcome: Phase 2: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) as of the 01 April 2011 Cut-off
Description: as for outcome 3
Time Frame: Up to week 70
Population: Safety population.
  Data collection is ongoing and future data results will be included as available.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2: Pomalidomide (Pom Only): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
  Data are reported during the time when participants were on pomalidomide alone, before dexamethasone was added.
- Phase 2: Pomalidomide (Pom + Dex Only): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
  Data are reported during the time after PD when participants were on both pomalidomide and dexamethasone.
- Phase 2: Pomalidomide (Overall): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing treatment or adding dexamethasone.
  Data are reported during the entire study up to the data cut-off, thus including both the time participants were only on pomalidomide and the time after PD when participants were on pomalidomide and dexamethasone.
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide (Pom Only) | Phase 2: Pomalidomide (Pom + Dex Only) | Phase 2: Pomalidomide (Overall)
Number analyzed (Participants) | 112 | 107 | 61 | 107
percentage of participants
  1 or more (1+) AE | 100.0 | 99.1 | 93.4 | 100.0
  1+ AE related to pomalidomide | 89.3 | 87.9 | 68.9 | 88.8
  1+ severity grade 3-4 AE | 88.4 | 84.1 | 70.5 | 89.7
  1+ severity grade 3-4 AE related to pomalidomide | 62.5 | 58.9 | 44.3 | 67.3
  1+ serious AE (SAE) | 61.6 | 46.7 | 47.5 | 67.3
  1+ SAE related to pomalidomide | 17.9 | 9.3 | 19.7 | 20.6
  1+ AE leading to discontinuation of pomalidomide | 8.0 | 10.3 | 3.3 | 12.1
  1+related AE --discontinuation of pomalidomide | 1.8 | 2.8 | 1.6 | 3.7
  1+AE - reduction of pomalidomide | 20.5 | 25.2 | 9.8 | 29.9
  1+ AE - interruption of pomalidomide | 63.4 | 47.7 | 36.1 | 58.9
  1+ related AE - interruption of pomalidomide | 27.7 | 24.3 | 21.3 | 32.7
  1+related AE - reduction of pomalidomide | 17.9 | 20.6 | 8.2 | 24.3

6. Secondary Outcome: Phase 2: Summary of Best Myeloma Response As Assessed by Independent Response Adjudication Committee (IRAC) Using European Group for Blood and Bone Marrow Transplant (EBMT) Criteria as of the 01 April 2011 Cut-off
Description: IRAC used EBMT criteria to assess myeloma response:
  * Complete Response (CR)-absence of serum and urine monoclonal paraprotein for 6 weeks, plus no increase in size or number of lytic bone lesions, plus other factors)
  * Partial Response (PR)-not all CR criteria, plus >=50% reduction in serum monoclonal paraprotein plus others
  * Minimal Response (MR)- 25-49% reduction in serum monoclonal paraprotein plus others
  * Stable Disease (SD)- not MR or progressive disease (PD)
  * Progressive Disease (PD)- reappearance of monoclonal paraprotein, lytic bone lesions, other
  * Not Evaluable (NE).
  Data collection is ongoing and future data results will be included as available.
Time Frame: up to 70 weeks
Population: Intent to treat population.
  Data collection is ongoing and future data results will be included as available.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2: Pomalidomide: 4 mg pomalidomide was given once per day on Days 1-21 of each 28-day cycle until PD. Participants in the single agent pomalidomide treatment arm who developed confirmed PD at any time had the option to receive oral dexamethasone at the starting dose in addition to their current dose of pomalidomide or to discontinue treatment.
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 113 | 108
percentage of participants
  Complete response (CR) | 0.9 | 0.0
  Partial response (PR) | 29.2 | 9.3
  Minimal response (MR) | 15.0 | 15.7
  Stable disease (SD) | 35.4 | 46.3
  Progressive disease (PD) | 6.2 | 15.7
  Not evaluable | 13.3 | 13.0

7. Secondary Outcome: Phase 2: Kaplan-Meier Estimates of Duration of Response as of the 01 April 2011 Cut-off
Description: Duration of myeloma response is defined as the time from when the response criteria are first met for partial response (PR) or better, until the first date the response criteria are met for progressive disease (PD) or until the participant dies from any cause, whichever occurs first. Duration of response for participants last known to be alive with no progression after a complete response (CR) or PR was censored at the date of last adequate response assessment. Participants with confirmed responses that occur after receiving any other anti-myeloma therapy (except for adding dexamethasone to the pomalidomide treatment arm), including radiation therapy initiated after baseline, was censored at the last adequate assessment prior to the initiation of such treatment.
  Response was assessed by the Independent Response Adjudication Committee (IRAC) using European Group for Blood and Bone Marrow Transplant (EBMT) criteria as described in the previous outcome.
Time Frame: up to 70 weeks
Population: Responders (participants with a complete response or partial response) from the ITT population.
  Data collection is ongoing and future data results will be included as available.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 34 | 10
weeks | 32.1 [22.1 to 39.9] | NA [NA to NA] — Not estimable since 9 or 10 responders were censored. The median was not reached at the time of the data cut-off.
Statistical Analysis 1: Comparison: Phase 2: Pomalidomide + Dexamethasone vs Phase 2: Pomalidomide; Test type: Superiority or Other; Cox Proportional Hazard = 6.25, 95% CI 2-sided [0.84 to 46.66]

8. Secondary Outcome: Phase 2: Time to Response as of the 01 April 2011 Cut-off
Description: Time to myeloma response is defined as the time from randomization to the time the response criteria for complete response (CR) or partial response (PR) are first met.
  Response was assessed by the Independent Response Adjudication Committee (IRAC) using European Group for Blood and Bone Marrow Transplant (EBMT) criteria as described previously.
  Data collection is ongoing and future data results will be included as available.
Time Frame: up to 70 weeks
Population: Responders (participants achieving CR or PR) from ITT population.
  Data collection is ongoing and future data results will be included as available.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 34 | 10
weeks | 8.1 [3.7 to 45.1] | 8.9 [4.1 to 49.6]
Statistical Analysis 1: Comparison: Phase 2: Pomalidomide + Dexamethasone vs Phase 2: Pomalidomide; Test type: Superiority or Other; p = 0.070, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Phase 2: Kaplan-Meier Estimates of Overall Survival as of the 01 April 2011 Cut-off
Description: Overall survival was defined as the time between randomization and death. Participants who die, regardless of the cause of the death, were considered to have had an event. All participants who were lost to follow-up prior to the end of the trial or who were withdrawn from the trial were censored at the time of last contact. Participants who were still being treated were censored at the last available date the subject was known to be alive, or clinical cut-off date if it was earlier.
  Data collection is ongoing and future data results will be included as available.
Time Frame: up to 70 weeks
Population: ITT population.
  Data collection is ongoing and future data results will be included as available.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 113 | 108
weeks | 62.6 [53.6 to NA] — Not estimable due to 69 out of 113 patients were still alive at data cutoff date | 59.3 [41.6 to NA] — Not estimable due to 61 out of 108 patients were still alive at data cutoff date
Statistical Analysis 1: Comparison: Phase 2: Pomalidomide + Dexamethasone vs Phase 2: Pomalidomide; Test type: Superiority or Other; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.57 to 1.29]

10. Primary Outcome: Phase 2: Percentage of Participants With Progression-Free Survival (PFS) Events as of the 01 April 2011 Cut-off
Description: Percentage of participants with the progression-free survival events: disease progression and death. Disease progression was assessed by the Independent Response Adjudication Committee (IRAC).
  Data collection is ongoing and future data results will be included as available.
Time Frame: up to 67 weeks
Population: Intent to treat population.
  Data collection is ongoing and future data results will be included as available.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide
Number analyzed (Participants) | 113 | 108
percentage of participants | 76.1 | 75.0

ADVERSE EVENTS:
Time Frame: Data cut-off 01 April 2011 Phase 1: up to 126 weeks Phase 2: up to 70 weeks
Groups:
- Phase 2: Pomalidomide (Pom Only): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing therapy or adding dexamethasone.
  Data are reported during the time when participants were on pomalidomide alone, before dexamethasone was added.
- Phase 2: Pomalidomide (Pom + Dex Only): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing therapy or adding dexamethasone.
  Data are reported during the time after PD when participants were on both pomalidomide and dexamethasone.
- Phase 2: Pomalidomide (Overall): Pomalidomide 4 mg daily on days 1-21 of each 28-day cycle. Upon PD, participants had the option of discontinuing therapy or adding dexamethasone.
  Data are reported during the entire study up to the data cut-off, thus including both the time participants were only on pomalidomide and the time after PD when participants were on pomalidomide and dexamethasone.
Arm/Group | Phase 1: 2 mg Pomalidomide | Phase 1: 3 mg Pomalidomide | Phase 1: 4 mg Pomalidomide | Phase 1: 5 mg Pomalidomide | Phase 2: Pomalidomide + Dexamethasone | Phase 2: Pomalidomide (Pom Only) | Phase 2: Pomalidomide (Pom + Dex Only) | Phase 2: Pomalidomide (Overall)
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/8 | 8/14 | 4/10 | 69/112 | 50/107 | 29/61 | 72/107
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 14/14 | 10/10 | 112/112 | 105/107 | 57/61 | 106/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 mg Pomalidomide (N=6) | Phase 1: 3 mg Pomalidomide (N=8) | Phase 1: 4 mg Pomalidomide (N=14) | Phase 1: 5 mg Pomalidomide (N=10) | Phase 2: Pomalidomide + Dexamethasone (N=112) | Phase 2: Pomalidomide (Pom Only) (N=107) | Phase 2: Pomalidomide (Pom + Dex Only) (N=61) | Phase 2: Pomalidomide (Overall) (N=107)
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 21 | 10 | 6 | 15
Sepsis (Infections and infestations) | 1 | 2 | 0 | 1 | 3 | 4 | 2 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Arthritis baterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 8 | 9 | 1 | 10
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 7 | 2 | 3 | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3 | 4 | 1 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 5
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 6 | 5 | 2 | 7
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 5
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardio-respiratory distress (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Brain mass (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Blood culture positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 mg Pomalidomide (N=6) | Phase 1: 3 mg Pomalidomide (N=8) | Phase 1: 4 mg Pomalidomide (N=14) | Phase 1: 5 mg Pomalidomide (N=10) | Phase 2: Pomalidomide + Dexamethasone (N=112) | Phase 2: Pomalidomide (Pom Only) (N=107) | Phase 2: Pomalidomide (Pom + Dex Only) (N=61) | Phase 2: Pomalidomide (Overall) (N=107)
Fatigue (General disorders) | 4 | 5 | 9 | 7 | 62 | 46 | 11 | 53
Pyrexia (General disorders) | 2 | 2 | 3 | 3 | 31 | 15 | 6 | 19
Oedema peripheral (General disorders) | 2 | 1 | 1 | 2 | 18 | 18 | 8 | 25
Asthenia (General disorders) | 3 | 2 | 1 | 0 | 22 | 11 | 5 | 15
Chills (General disorders) | 1 | 0 | 1 | 1 | 12 | 9 | 2 | 10
Malaise (General disorders) | 0 | 2 | 2 | 3 | 4 | 5 | 1 | 6
Gait disturbance (General disorders) | 1 | 0 | 1 | 1 | 4 | 6 | 3 | 8
Pain (General disorders) | 0 | 0 | 1 | 0 | 5 | 5 | 1 | 6
Irritability (General disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 8 | 9 | 52 | 53 | 17 | 55
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 5 | 3 | 43 | 36 | 11 | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 3 | 24 | 25 | 7 | 27
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 19 | 11 | 2 | 12
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 17 | 4 | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 4 | 38 | 29 | 11 | 38
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 37 | 22 | 17 | 35
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 5 | 24 | 29 | 10 | 37
Vomiting (Gastrointestinal disorders) | 1 | 2 | 4 | 2 | 15 | 10 | 4 | 14
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 8 | 9 | 0 | 9
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 5 | 5 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 8 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 4 | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 1 | 32 | 26 | 10 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 2 | 21 | 17 | 7 | 20
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 21 | 16 | 8 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 17 | 14 | 3 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 17 | 8 | 4 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 12 | 8 | 5 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 15 | 4 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 5 | 7 | 6 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 5 | 4 | 2 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2 | 3 | 33 | 23 | 6 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 2 | 23 | 14 | 4 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 12 | 12 | 4 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 17 | 9 | 4 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 11 | 4 | 2 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 10 | 7 | 1 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 7 | 4 | 3 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 4 | 3 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 7 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 5 | 2 | 23 | 17 | 10 | 27
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 1 | 15 | 7 | 2 | 8
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 8 | 6 | 5 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 4 | 2 | 4 | 6
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 2 | 5 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 4 | 1 | 5
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 6 | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 3
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Urethritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 3 | 19 | 15 | 8 | 23
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 11 | 17 | 3 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 17 | 10 | 4 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 14 | 7 | 3 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 12 | 6 | 5 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 13 | 5 | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 5 | 4 | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 7 | 4 | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 9 | 4 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 4 | 7 | 0 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 5 | 4 | 2 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 8 | 2 | 1 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 18 | 22 | 2 | 23
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 18 | 4 | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 8 | 14 | 1 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 12 | 9 | 1 | 10
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 14 | 3 | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 2 | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ingrown nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichenoid karatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 4 | 2 | 19 | 16 | 4 | 20
Headache (Nervous system disorders) | 0 | 0 | 3 | 2 | 9 | 12 | 2 | 14
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 14 | 7 | 3 | 10
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 3 | 8 | 11 | 0 | 11
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 4 | 4 | 2 | 5
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 6 | 3 | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 8 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 4 | 2 | 6
Numb chin syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 12 | 11 | 6 | 14
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 9 | 9 | 5 | 15
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 12 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 7 | 5 | 0 | 5
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 8 | 5 | 1 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 2
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 1 | 16 | 0 | 7 | 7
Confusional state (Psychiatric disorders) | 1 | 2 | 1 | 0 | 14 | 6 | 3 | 9
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 0 | 8 | 9 | 3 | 12
Depression (Psychiatric disorders) | 0 | 0 | 3 | 2 | 3 | 3 | 3 | 6
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 2
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 2 | 3 | 9 | 4 | 0 | 4
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 3 | 3 | 1 | 4
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Eyelid disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 6 | 5 | 1 | 6
Hot flush (Vascular disorders) | 0 | 1 | 1 | 0 | 5 | 3 | 1 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 5 | 1 | 2 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 4 | 3 | 5
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 6
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 3 | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 9 | 3 | 1 | 4
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic oedema (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, and has priority over subset (single center) publication, for 1 year after study completion.
* Investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. Celgene has 45 days to review and comment on draft manuscript/presentation, and may ask for an additional delay (not to exceed 90 days total) to address intellectual property issues.